CLINICAL TRIAL: NCT02933346
Title: Assessment and Follow-up of Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Nivolumab Under the French Temporary Authorization for Use (ATU) Program
Brief Title: Cohort of Patients With NSCLC Treated With Nivolumab Under the ATU Program
Acronym: CLINIVO
Status: Completed | Type: Observational
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IFCT-1502 CLINIVO
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Non-small Cell Lung Cancer; Nivolumab; Long-term Adverse Effects
Keywords: Nivolumab; Real-world study; IFCT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Long Term Adverse Effects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Our study sought to examine nivolumab efficacy and safety in advanced NSCLC patients treated under the Temporary Authorization for Use (ATU, compassionate use) setting and describe their long-term clinical characteristics, notably the treatments they received after nivolumab discontinuation. The profile of these patients shows greater conformity to that of a non-selected population, yet the clinical data collection does not reflect "real life" conditions and stops when treatment ends, which does not enable us to get an overview of post-immunotherapy treatments.

DETAILED DESCRIPTION:
Although the oncogene addiction concept has led to effective targeted treatments for certain histological non-small cell lung cancer (NSCLC) types, most patients with advanced tumors are still treated with first-line chemotherapy. In 2015, several studiess demonstrated the efficacy of nivolumab, an immunotherapy targeting immune checkpoints. In France, besides the clinical trials, this molecule has been made available in January 2015 under a Temporary Authorization for Use (ATU, compassionate use).

Our study sought to examine nivolumab efficacy and safety in advanced NSCLC patients treated under the ATU setting and describe their long-term clinical characteristics, notably the treatments they received after nivolumab discontinuation. The profile of these patients shows greater conformity to that of a non-selected population, yet the clinical data collection does not reflect "real life" conditions and stops when treatment ends, which does not enable us to get an overview of post-immunotherapy treatments.

ELIGIBILITY:
Inclusion Criteria:

* All patients with advanced NSCLC, non-eligible for thoracic radiation therapy, having received nivolumab (at least one injection), under nominative or cohort ATU, between 23-JAN-2015 and 31-AUG-2015 (end of ATU).

Exclusion Criteria:

* patients included in a biomedical research trial with nivolumab
* patients <18 years old
* patients included under ATU to receive nivolumab administration, but never did
* patients with a psychiatric history that hinders the comprehension of the information leaflet
* patients refusing their data being collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with advanced NSCLC, non-eligible for thoracic radiation therapy, having received nivolumab (at least one injection), under nominative or cohort ATU, between 23-JAN-2015 and 31-AUG-2015 (end of ATU).
Sampling Method: Non-Probability Sample
Enrollment: 907 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
overall survival | January 2015 - December 2017
  time from start of treatment to death from any cause

SECONDARY OUTCOMES:
efficacy of nivolumab | January 2015 - December 2017
  progression-free survival, best overall response, exposure time
maximum toxicities of nivolumab treatment, including delayed toxicities (immune) | January 2015 - December 2017
  Maximum toxicity according to the investigator (Adverse events with NCI-CTC 4.0 Grade ≥2, categorized as: hepatic, pulmonary, endocrine, cutaneous, gastrointestinal, renal, hematologic, other immune toxicities)
efficacy of the first systemic treatment post-nivolumab | January 2015 - December 2017
  progression-free survival, best response

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MOLINIER, MD, Principal Investigator — CH Le Mans, France
Locations (72):
- France (72):
  - CH du Pays d'Aix, Aix-en-Provence
  - Clinique du Rambot, Aix-en-Provence
  - CHU d'Amiens-Picardie, Amiens
  - CHU d'Angers, Angers
  - CH Argenteuil, Argenteuil
  - CH d'Avignon, Avignon
  - Institut Sainte Catherine, Avignon
  - CH de la Côte Basque, Bayonne
  - CHU de Besançon, Besançon
  - CH de Blois, Blois
  - Hôpital Avicenne APHP, Bobigny
  - CH Briançon, Briançon
  - Hôpital Pradel HCL, Bron
  - Caen CLCC, Caen
  - CHU de Caen, Caen
  - CH de Pontoise, Cergy-Pontoise
  - CH Métropole Savoie, Chambéry
  - HIA Percy, Clamart
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CH Alpes Léman, Contamine-sur-Arve
  - Clinique des Cèdres, Cornebarrieu
  - CHI de Créteil, Créteil
  - CH de Dax, Dax
  - Centre Georges-François Leclerc, Dijon
  - Institut Daniel Hollard, Grenoble
  - CHR Saint-Omer, Helfaut
  - CHD Vendée, La Roche-sur-Yon
  - CHU Grenoble Alpes, La Tronche
  - CH de Versailles, Le Chesnay
  - Hôpital Bicêtre APHP, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - CHRU de Lille, Lille
  - CHU de Limoges, Limoges
  - Polyclinique de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - HP Clairval, Marseille
  - Hôpital Nord APHM, Marseille
  - HP Robert Schumann, Metz
  - CH de Mont-De-Masan, Mont-de-Marsan
  - CH de Belfort Montbéliard, Montbéliard
  - GRH Mulhouse Sud-Alsace, Mulhouse
  - Centre d'Oncologie de Gentilly, Nancy
  - Nice CLCC, Nice
  - CHU Nîmes, Nîmes
  - CHR d'Orléans, Orléans
  - Hegp Aphp, Paris
  - HIA Val de Grâce, Paris
  - Hôpital Saint Joseph, Paris
  - Hôpital Saint Louis APHP, Paris
  - Hôpital Tenon APHP, Paris
  - CH de Pau, Pau
  - CHU de Bordeaux, Pessac
  - CH Lyon-Sud HCL, Pierre-Bénite
  - CH de Saint-Brieuc, Saint-Brieuc
  - CHU de Nantes, Saint-Herblain
  - ICO René Gauducheau, Saint-Herblain
  - CH Annecy Genevois, Saint-Julien-en-Genevois
  - HIA Begin, Saint-Mandé
  - ICL Lucien Neuwirth, Saint-Priest-en-Jarez
  - NHC CHRU de Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes
  - CHI Toulon La Seyne Sur Mer, Toulon
  - HIA Saint Anne, Toulon
  - CHU Toulouse, Toulouse
  - CHRU de Tours, Tours
  - Clinique Saint Joseph, Trélazé
  - CH de Valence, Valence
  - CHU Bretagne Atlantique, Vannes
  - Hôpital Nord-Ouest, Villefranche-sur-Saône
  - Gustave Roussy, Villejuif
  - Hôpital Paul Brousse APHP, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Molinier O, Besse B, Barlesi F, Audigier-Valette C, Friard S, Monnet I, Jeannin G, Mazieres J, Cadranel J, Hureaux J, Hilgers W, Quoix E, Coudert B, Moro-Sibilot D, Fauchon E, Westeel V, Brun P, Langlais A, Morin F, Souquet PJ, Girard N. IFCT-1502 CLINIVO: real-world evidence of long-term survival with nivolumab in a nationwide cohort of patients with advanced non-small-cell lung cancer. ESMO Open. 2022 Feb;7(1):100353. doi: 10.1016/j.esmoop.2021.100353. Epub 2021 Dec 23. PMID 34953398